CLINICAL TRIAL: NCT00148239
Title: Caregiver Intervention for Caregivers of SCI Patients
Brief Title: Health Interventions for Survivors and Primary Support Persons of Spinal Cord Injury
Acronym: SCI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, Richard Schulz, Prof. of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01NR008272 (NIH)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Cord Injuries
Keywords: SCI; Caregiving; Aging; Disability; Paralysis
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Caregiver Only (Experimental): A multi-component psycho-educational intervention designed to reduce the negative emotional and behavioral responses of the caregiver and reduce the risk of mental and physical health problems.
  Interventions: Behavioral: Caregiver Only Intervention
- Dual Treatment (Experimental): Complements the caregiver only intervention by targetting both caregiver and SCI person with multi-component psycho-educational intervention
  Interventions: Behavioral: Dual Treatment
- Control (Active Comparator): Participants are provided with written materials at beginning of study; nothing thereafter
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Caregiver Only Intervention — A multi-component psycho-educational intervention designed to reduce the negative emotional and behavioral responses of the caregiver and reduce the risk of mental and physical health problems.
  Arms: Caregiver Only
Behavioral: Dual Treatment — Complements the caregiver only intervention by targetting both caregiver and SCI person with multi-component psycho-educational intervention
  Arms: Dual Treatment
Behavioral: Control — Participants given written educational materials at beginning of study; no treatment beyond this
  Arms: Control

SUMMARY:
The overall objective of this project is to test the efficacy of an innovative multi-component intervention aimed at reducing the risk for adverse health outcomes among caregivers of older survivors with spinal cord injury or disability, and to improve the well being of the spinal cord-injured survivor. In a three-group, randomized, controlled design providing access to information, resources, and support, we predict that the dual target approach will have a greater positive impact on both the caregiver and survivor than the caregiver-only approach, and that both active treatments will be superior with respect to caregiver outcomes than an information-only control condition.

DETAILED DESCRIPTION:
The specific aims of this project are to:

1. Assess the impact of a dual target (caregiver and care recipient) intervention compared to a traditional caregiver-only intervention strategy.
2. Assess causal linkages between the treatment components (e.g. knowledge, social support) of a multi-component intervention and specific treatment outcomes (e.g. caregiver depression, quality of life).
3. Explore cultural and racial differences in the evaluation of and effectiveness of the different treatment approaches.

Overall, the issues affecting management of SCI/D in later life are complex and hold critical implications for the health of the long-term survivor as well as for those who provide care in the home environment. Large numbers of individuals are living with the effects of SCI/D for decades post-injury. In addition to the health-related complications that typically accompany older age, these individuals are especially vulnerable to co-occurring medical conditions that require high degrees of support and maintenance. Consequently, older caregivers face multiple and often extreme challenges in providing support to the SCI/D survivor at a time in their lives when their own abilities may be compromised due to age-related changes in health and functioning.

The multi-faceted burden faced by caregivers is associated with high levels of depression and anxiety as well as the onset of deleterious physical symptoms. The cumulative effects of such multiple stressors over time all too frequently leave the caregiver unable to continue providing the level of support necessary to maintain their partner's health in the home environment. In order to circumvent the additional distress certain to accompany such a family separation, Elliott et al. (2001, p. 230) recently concluded that "there is a pressing need for interventions that help family [SCI] caregivers address the routines and tasks essential to maintaining family functioning."

ELIGIBILITY:
Inclusion Criteria (Survivors):

* have adult-onset disability resulting from spinal cord injury, trauma, or disease,
* be survivors with complete or incomplete injury as defined by the American Spinal Injury Association (ASIA) impairment scale
* require and use some type of assistance for getting around (e.g., wheelchair, cane, etc.) be 30 years old or older be living at home for a minimum of 1 year post-injury (to avoid the acute trauma phase) speak English.

Inclusion Criteria (Caregivers):

* Is a family member/partner (e.g. spouse, child, or fictive kin)
* is 18 years of age or older
* is or is not living with the care recipient
* speaks English
* has a telephone at home
* plans to live in the area for at least 6 months.
* self-identifies as white, African American or Hispanic.

Exclusion Criteria:

* has a terminal illness with life expectancy of less than 6 months
* is in active treatment for cancer (except for tamoxifen and lupron)
* is blind or deaf
* if the survivor is cognitively impaired due to brain injury or dementia and/or has no use of their hands and severe limitations in speech production

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2002-09; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms caregivers and SCI | 6 and 12 months post-randomization
Caregiver Burden | 6 and 12 months
Social support caregiver and SCI | 6 and 12 months
Health symptoms caregiver and SCI | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schulz, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - University of Pittsburgh (UCSUR), Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Schulz R, Czaja SJ, Lustig A, Zdaniuk B, Martire LM, Perdomo D. Improving the quality of life of caregivers of persons with spinal cord injury: a randomized controlled trial. Rehabil Psychol. 2009 Feb;54(1):1-15. doi: 10.1037/a0014932. PMID 19618698